CLINICAL TRIAL: NCT03639857
Title: A Comparative Study of the Efficacy of 532nm Laser and 1064 nm Laser in the Treatment of Cutaneous Lupus Erythematous Versus Topical Corticosteroids Alone
Brief Title: Study of the Efficacy of 532nm Laser and 1064 nm Laser in the Treatment of Cutaneous Lupus Erythematous Versus Topical Corticosteroids Alone
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Time and resource constraints
Sponsor: David Weinstein (Other)
Responsible Party: Sponsor-Investigator, David Weinstein, Assistant Professor of Dermatology, University of Central Florida
Organization: University of Central Florida (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BIO-17-13680
Record Dates: First submitted 2018-08-17; First posted 2018-08-21 (Actual); Results first posted 2021-07-21 (Actual); Last update posted 2021-07-21 (Actual); Status verified 2021-06

CONDITIONS: Cutaneous Lupus
MeSH Terms: interventions — Lasers; Adrenal Cortex Hormones

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (3):
- 532nm laser and topical corticosteroid (Experimental): 532nm laser is applied to the patient's lesion in-clinic in addition to a topical corticosteroid.
  Interventions: Device: 532nm laser; Drug: Topical corticosteroid
- 1064nm laser and topical corticosteroid (Experimental): 1064nm laser is applied to the patient's lesion in-clinic in addition to a topical corticosteroid.
  Interventions: Device: 1064nm laser; Drug: Topical corticosteroid
- Topical corticosteroid alone (Active Comparator): Topical corticosteroid is applied to the patient's lesion.
  Interventions: Drug: Topical corticosteroid

INTERVENTIONS:
Device: 532nm laser — 532nm laser will be used to treat the lesion in this study arm.
  Arms: 532nm laser and topical corticosteroid
Device: 1064nm laser — 1064nm laser will be used to treat the lesion in this study arm.
  Arms: 1064nm laser and topical corticosteroid
Drug: Topical corticosteroid — The topical corticosteroid will be used to treat the lesion in this study arm.

SUMMARY:
This study aims to compare the efficacy of 532nm Potassium Titanyl Phosphate (KTP) laser and 1064 nm Neodymium-doped Yttrium Aluminum Garnet (Nd:YAG) laser as adjuncts to topical corticosteroids in the treatment of cutaneous lupus erythematosus versus topical corticosteroids alone.

ELIGIBILITY:
Inclusion Criteria:

* Male or female adult 18 years of age or older
* Ability to rate level of pain
* Ability to rate visual satisfaction
* At least 2 active lesions of CLE

Exclusion Criteria:

* New or change in systemic medication for cutaneous lupus in past 6 months
* Allergy to triamcinolone or betamethasone dipropionate cream
* Pregnancy
* Currently a prisoner
* Unable to read and speak English since consent will only be available in English

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2018-08-17 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- UCF Health Lake Nona Office, Orlando, Florida, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: We had planned to enroll 7 participants but due to lack of resources/support the study ended early with only 3 participants.
Units Other Than Participants: Lesions
Period: Overall Study
Arm/Group | 532nm Laser and Topical Corticosteroid | 1064nm Laser and Topical Corticosteroid | Topical Corticosteroid Alone
Started | 1; 1 Lesions | 3; 3 Lesions | 3; 3 Lesions
Completed | 1; 1 Lesions | 3; 3 Lesions | 3; 3 Lesions
Not Completed | 0; 0 Lesions | 0; 0 Lesions | 0; 0 Lesions

BASELINE CHARACTERISTICS:
Units Other Than Participants: Lesions
Groups:
- All Study Participants: All study participants received treatment of 2 or 3 lesions of cutaneous lupus depending upon their skin type.
  Participants with skin type 1, 2 or 3 received treatment of 3 lesions:
  * One lesion treated with 532nm laser
  * One lesion treated with the 1064nm laser
  * One lesion treated with topical corticosteroid
  Participants with skin type 4, 5 or 6 received treatment of 2 lesions
  * One lesion treated with the 1064nm laser
  * One lesion treated with topical corticosteroid
Arm/Group | All Study Participants
Number analyzed (Participants) | 3
Number analyzed (Lesions) | 7
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 3
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
  Participants
    number analyzed (Participants) | 0
Region of Enrollment [Number; unit: participants]
  United States | 3

OUTCOME MEASURES:

1. Primary Outcome: Limited CLASI
Description: The investigators are using a limited Cutaneous Lupus Erythematosus Disease Area and Severity Index (CLASI) scoring system to classify specific lesions the investigators are measuring. The total limited CLASI reflects the sum of both active and damage CLASI, resulting in a score ranging from 0 to 8. A higher score indicates more severe disease. Score is assessed by the investigators.
  The limited active CLASI for a lesion will include the following:
  * Erythema (ranging from 0 = absent to 3 = dark red/purple)
  * Scale/Hypertrophy (ranging from 0 = absent to 2 = verrucous/ hypertrophic)
  * The addition of these scores result in a total limited active CLASI score of the studied lesion, ranging from 0 to 5.
  The limited damage CLASI for a lesion will include the following:
  * Dyspigmentation (0 = absent or 1 = present)
  * Scarring/Atrophy/Panniculitis (ranging from 0 = absent to 2 = severely atrophic scarring or panniculitis).
  * The addition of these scores result in a
Time Frame: 2 Months
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | 532nm Laser and Topical Corticosteroid | 1064nm Laser and Topical Corticosteroid | Topical Corticosteroid Alone
Number analyzed (Participants) | 1 | 3 | 3
score on a scale
  Baseline | 5 [5 to 5] | 4 [2 to 5] | 4.3 [3 to 6]
  1 Month | 5 [5 to 5] | 3.66 [2 to 5] | 4 [3 to 5]
  2 Months | 5 [5 to 5] | 3.66 [2 to 6] | 4.33 [3 to 6]

2. Primary Outcome: VAS for Appearance
Description: The investigators are using a VAS (visual analog scale) to measure patient assessment of the appearance of the lesion. The scale ranges from 0-10, with 10 being very satisfied and 0 being no satisfaction at all.
  A score of 0 will represent a cosmetically fully unsatisfactory result and 10 will represent cosmetically excellent result.
Time Frame: 2 Months
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | 532nm Laser and Topical Corticosteroid | 1064nm Laser and Topical Corticosteroid | Topical Corticosteroid Alone
Number analyzed (Participants) | 1 | 3 | 3
score on a scale
  Baseline | 7.5 [7.5 to 7.5] | 3.2 [1.4 to 6.3] | 4.2 [1.8 to 5.5]
  1 Month | 10 [10 to 10] | 7.5 [6.4 to 9] | 5.5 [3.5 to 8]
  2 Months | 9 [9 to 9] | 6.5 [4 to 7.8] | 3.6 [2 to 5.5]

3. Primary Outcome: VAS for Pain
Description: The investigators are using a VAS (visual analog scale) to assess pain of the laser treatment. The participant rates the pain of the laser treatment. The scale ranges from 0 (no pain) to 10(worse pain).
  A score of 0 will represent absence of pain and 10 will represent maximal pain.
Time Frame: 1 Month
Population: The control arm did not receive any laser intervention, just a topical medication therefore the pain scale was not used.
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | 532nm Laser and Topical Corticosteroid | 1064nm Laser and Topical Corticosteroid | Topical Corticosteroid Alone
Number analyzed (Participants) | 1 | 3 | 0
score on a scale
  Baseline | 1.4 [1.4 to 1.4] | 3.1 [0 to 5] |
  1 Month | 6 [6 to 6] | 2.13 [1 to 3.1] |

ADVERSE EVENTS:
Time Frame: Adverse Events and All-Cause Mortality were assessed for 8 weeks of treatment and 1 month after for follow-up.
Description: This was only a moderate risk study for the participants as only a lower energy laser was used on the skin.
Arm/Group | 532nm Laser and Topical Corticosteroid | 1064nm Laser and Topical Corticosteroid | Topical Corticosteroid Alone
All-Cause Mortality (participants affected / at risk) | 0/1 | 0/3 | 0/3
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/3 | 0/3
Other Adverse Events (participants affected / at risk) | 0/1 | 0/3 | 0/3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-05-22): https://cdn.clinicaltrials.gov/large-docs/57/NCT03639857/Prot_SAP_002.pdf
  • Informed Consent Form (2019-05-22): https://cdn.clinicaltrials.gov/large-docs/57/NCT03639857/ICF_003.pdf